CLINICAL TRIAL: NCT06028191
Title: Combined Effects of Low Level Laser Therapy and Kabat Technique in Patients With Bell's Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0229
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Bell Palsy
Keywords: Bell's Palsy; Facial Disability Index; Kabat Technique; Low Level Laser Therapy; Sunnybrook facial grading system
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kabat Technique along with baseline treatment (Other): Kabat technique will be performed for 15 min along with baseline treatment will be given to Group A. They will have 45 min-1 hour session thrice a week in duration of six weeks.
  Interventions: Other: Kabat Technique along with baseline treatment
- Kabat Technique and LLLT along with baseline treatment (Experimental): Kabat technique will be performed for 15 min and LLLT will be performed for 10 min to eight points of the effected side for 2 min at each point along with baseline treatment. They will have 45 min-1 hour session thrice a week in duration of six weeks
  Interventions: Device: Kabat Technique and LLLT along with baseline treatment

INTERVENTIONS:
Other: Kabat Technique along with baseline treatment — Group A will receive Kabat Technique along with baseline treatment. Electrical muscle stimulation for 15 min which includes faradic current to the facial nerve trunks given by DL-2 electro pulse stimulator, Effleurage and Kneading for 5 min and resistive exercise for 5 min and facial expression exercises for 5 min, which included eye closure, eyebrow raise, frown, smile, snarl, pucker and pout as baseline treatment.
  Kabat Technique is neurorehabilitation technique that uses diagonal and spiralpatterns for movement in conjunction with stretch and resistance and other PNF techniques to reinforce neuromuscular recruitment. It mainly concerns the stimulation of these muscles: Orbicularis occuli, ztgomaticus, Levator labii, nasalis, buccinator, frontalis, corrugator
  Other Names: Group A
  Arms: Kabat Technique along with baseline treatment
Device: Kabat Technique and LLLT along with baseline treatment — Group B will receive Kabat Technique and LLLT along with baselinetreatment. Kabat technique is same as mentioned in group A. Laser treatment will be administered to eight points of the affected side for 2 min at each point at a wavelength of 830 nm, output power of 100 Mw, and frequency of 1 KHz. Endo laser 422 is the model name and number of device which will be used in this study to administered low level laser therapy.
  Other Names: Group B
  Arms: Kabat Technique and LLLT along with baseline treatment

SUMMARY:
The objective of this current study is to determine the combined effects of Low-Level Laser Therapy (LLLT) and the Kabat technique on quality of life, synkinetic movements and functional outcome in patients of Bell's palsy

DETAILED DESCRIPTION:
Bell's palsy is an acute condition which occurs by the damage of 7th cranial nerve along its course at the level which is distal to Pons. Basically it is an idiopathic facial condition.

The yearly incidence of Bell's palsy is 15 to 30 per 100,000 people, which affect both sexes equally. This study aims to see combined effects of Low Level Laser Therapy and Kabat technique in the treatment of Bell's palsy.

Synkinesis, which is described as an involuntary movement in one part of the face produced during voluntary movement in another region of the face, is a problematic Bell's palsy sequel. The mechanism behind the formation of synkinesis is unknown. According to the predominant idea, damaged axons regenerate abnormally, innervating facial muscles that weren't originally innervated. The yearly incidence of Bell's palsy is 15 to 30 per 100,000 people, which affect both sexes equally.

Kabat Technique is neurorehabilitation technique that uses diagonal and spiral patterns for movement in conjunction with stretch and resistance and other PNF techniques to reinforce neuromuscular recruitment. It mainly concerns the stimulation of these muscles: Orbicularis occuli, ztgomaticus, Levator labii, nasalis, buccinator, frontalis, corrugator.

For all BP patients, including those who are unable to take corticosteroids due to diabetes or hypertension, laser therapy offers a non-invasive, painless means of treatment. However, just a few researches have examined the effectiveness of low- dose laser therapy in BP patients.

Low Level Laser Therapy has the potential to promote nerve regeneration, reduce inflammation, and accelerate tissue healing in the affected facial nerve. On the other hand, the Kabat technique focuses on restoring neuromuscular control and improving muscle function. By combining Low Level Laser Therapy and the Kabat technique, a synergistic effect may be achieved, maximizing the potential benefits of both interventions. Therefore, this study aims to determine the specific parameters and protocols for the combined use of Low Level Laser Therapy and the Kabat technique in Bell's palsy

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Both genders will be included
* Unilateral Facial paralysis/paresis
* Patients presented within onset of 12 days - 3 weeks (sub-acute Bell's Palsy)

Exclusion Criteria:

* Previous surgery of facial reconstruction
* Traumatic Brain Injury
* Any other neurological deficit
* Congenital Deformities
* Recurrent Bell's palsy will be excluded

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Sunnybrook Facial Grading system | 6 weeks
  Sunnybrook facial grading system was used to quantify the symmetry of voluntary and resting muscles

SECONDARY OUTCOMES:
Facial disability index | 6 weeks
  it has two components. The physical function subscale detects problems in drinking, speaking eating, lacrimation, and oral hygiene. The social/well-being function subscale detects subjective irritation, perception of anxiety, and isolation; problems in sleeping; and limitations in social participation.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Tariq, Mphil, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Allied Hospital, Faisalābad, Punjab Province
  - Physiofit, Faisalābad, Punjab Province

IPD SHARING:
Plan to Share IPD: No